CLINICAL TRIAL: NCT00667342
Title: A Study of Bevacizumab, a Humanized Monoclonal Antibody Against Vascular Endothelial Growth Factor (VEGF), in Combination With Chemotherapy for Treatment of Osteosarcoma
Brief Title: A Study of Bevacizumab in Combination With Chemotherapy for Treatment of Osteosarcoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: St. Jude Children's Research Hospital (Other)
Collaborators: Genentech, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: OS2008; GENENTECH PHARM (Other: Genentech Pharmaceuticals); NCI-2009-00846 (Registry Identifier: NCI Clinical Trial Registration Program)
Record Dates: First submitted 2008-04-24; First posted 2008-04-28 (Estimated); Results first posted 2014-08-04 (Estimated); Last update posted 2023-08-07 (Actual); Status verified 2019-05

CONDITIONS: Osteosarcoma; Malignant Fibrous Histiocytoma (MFH) of Bone
MeSH Terms: conditions — Osteosarcoma; Histiocytoma, Malignant Fibrous | interventions — Bevacizumab; Cisplatin; Doxorubicin; Methotrexate; Ifosfamide; Etoposide; Surgical Procedures, Operative; Radiotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Localized Resectable Disease (Stratum A) (Experimental): Participants with localized resectable disease receive Cycle 1 of bevacizumab 3 days before chemotherapy with cisplatin and doxorubicin. Subsequent cycles consist of bevacizumab on the first day of chemotherapy, then cisplatin, and doxorubicin, or methotrexate. If applicable, definitive surgery and assessment of histologic response will occur at week 10 followed by bevacizumab on the first day of chemotherapy with cisplatin and doxorubicin, or methotrexate.
  Interventions: Biological: Bevacizumab; Drug: Cisplatin; Drug: Doxorubicin; Drug: Methotrexate; Procedure: Surgery
- Metastatic Disease (Stratum B) (Experimental): Participants with metastatic disease (Stratum B) receive Cycle 1 of bevacizumab 3 days before chemotherapy with cisplatin and doxorubicin. Subsequent cycles consist of bevacizumab on the first day of chemotherapy, then cisplatin and doxorubicin, methotrexate or ifosfamide, and etoposide. If applicable, definitive surgery and assessment of histologic response will occur at week 10 followed by bevacizumab on the first day of chemotherapy with cisplatin and doxorubicin, methotrexate, or ifosfamide, and etoposide. Radiotherapy will be given post-operatively.
  Interventions: Biological: Bevacizumab; Drug: Cisplatin; Drug: Doxorubicin; Drug: Methotrexate; Drug: Ifosfamide; Drug: etoposide; Procedure: Surgery; Radiation: Radiotherapy
- Unresectable Disease (Stratum C) (Experimental): Participants with unresectable disease (Stratum C) receive treatment identical to Stratum B: Cycle 1 of bevacizumab 3 days before chemotherapy with cisplatin and doxorubicin. Subsequent cycles consist of bevacizumab on the first day of chemotherapy, then cisplatin and doxorubicin, methotrexate or ifosfamide, and etoposide. If applicable, definitive surgery and assessment of histologic response will occur at week 10 followed by bevacizumab on the first day of chemotherapy with cisplatin and doxorubicin, methotrexate, or ifosfamide, and etoposide. Radiotherapy will be given post-operatively.
  Interventions: Biological: Bevacizumab; Drug: Cisplatin; Drug: Doxorubicin; Drug: Methotrexate; Drug: Ifosfamide; Drug: etoposide; Procedure: Surgery; Radiation: Radiotherapy

INTERVENTIONS:
Biological: Bevacizumab — Monoclonal Antibody against vascular endothelial growth factor (VEGF). Given intravenously (IV).
  Other Names: rhuMAb VEGF; Avastin®
Drug: Cisplatin — Given IV.
  Other Names: Platinol-AQ®
Drug: Doxorubicin — Given IV.
  Other Names: Adriamycin®
Drug: Methotrexate — Given IV.
  Other Names: MTX
Drug: Ifosfamide — Given IV.
  Other Names: Ifex®
  Arms: Metastatic Disease (Stratum B); Unresectable Disease (Stratum C)
Drug: etoposide — Given IV.
  Other Names: VP-16; Vepesid®
  Arms: Metastatic Disease (Stratum B); Unresectable Disease (Stratum C)
Procedure: Surgery — Participants undergo definitive surgery and assessment of histologic response at week 10.
Radiation: Radiotherapy — Radiation therapy delivered for positive margins or intralesional resections.
  Arms: Metastatic Disease (Stratum B); Unresectable Disease (Stratum C)

SUMMARY:
This study adopts a novel strategy for first-line treatment of osteosarcoma by combining chemotherapy with anti-angiogenic therapy using bevacizumab (Avastin®), a humanized monoclonal antibody against vascular endothelial growth factor (VEGF). Chemotherapy for localized disease comprises a 3-drug regimen (cisplatin, doxorubicin, and high-dose methotrexate). Chemotherapy for metastatic or unresectable disease comprises a cisplatin-based regimen that includes high-dose methotrexate, doxorubicin, ifosfamide, and etoposide.

DETAILED DESCRIPTION:
This is a comprehensive study that uses a novel agent that targets angiogenesis (bevacizumab) in combination with conventional chemotherapy for the treatment of osteosarcoma. Bevacizumab, a monoclonal antibody against the vascular endothelial growth factor (VEGF), has been shown to stop the growth of new blood vessels of tumors, both in the laboratory and in patients with other types of cancers. Bevacizumab has improved the effect of chemotherapy in adult patients with different types of cancer by increasing tumor response and increasing the chances of survival. This study has two main goals:

* To find out if bevacizumab can be combined safely with chemotherapy for osteosarcoma
* To find out if adding bevacizumab to chemotherapy will be beneficial in treating osteosarcoma.

The chemotherapy drugs used in this study are commonly used to treat osteosarcoma. Patients with non-metastatic and resectable tumors receive bevacizumab and chemotherapy comprised of cisplatin, doxorubicin and high-dose methotrexate. Patients with metastatic tumors or tumors that cannot be removed by surgery receive bevacizumab and chemotherapy comprised of cisplatin, doxorubicin and high-dose methotrexate, ifosfamide and etoposide. If the tumor can be removed by surgery, surgery will be performed after 10 weeks of chemotherapy and will be followed by additional chemotherapy. After completion of active therapy, patient's response to therapy will be followed for approximately 5 years.

ELIGIBILITY:
Inclusion Criteria:

* Patient must have newly diagnosed high-grade, biopsy proven, osteosarcoma or malignant fibrous histiocytoma (MFH) of bone with no history of prior chemotherapy or radiation;
* Participant is able to perform tasks and daily activities as defined in the study guidelines
* Patient meets established guidelines for adequate function of the kidney, liver, heart and bone marrow
* Participants meets other requirements defined in the eligibility portion of the study

Exclusion Criteria:

* recent major surgical procedure or injury
* Known bleeding diathesis, platelet disorder or coagulopathy
* Thrombosis
* Cardiac disease or hypertension
* Significant proteinuria
* Central nervous system disease
* Gastrointestinal perforation/abdominal fistula
* Osteosarcoma or MFH of bone as second malignancy

Max Age: 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 43 (Actual)
Dates: Start 2008-06-03 (Actual); Primary Completion 2014-08 (Actual); Study Completion 2017-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Michael Bishop, MD, Principal Investigator — St. Jude Children's Research Hospital
Locations (5):
- United States (5):
  - Rady Children's Hospital and Health Center, San Diego, California
  - Johns Hopkins - Sidney Kimmel Comprehensive Cancer Center, Baltimore, Maryland
  - NCI/NIH - Pediatric Oncology Branch, Bethesda, Maryland
  - St Jude Children's Research Hospital, Memphis, Tennessee
  - MD Anderson Cancer Center, Houston, Texas

REFERENCES:
- [Derived] Turner DC, Navid F, Daw NC, Mao S, Wu J, Santana VM, Neel M, Rao B, Willert JR, Loeb DM, Harstead KE, Throm SL, Freeman BB 3rd, Stewart CF. Population pharmacokinetics of bevacizumab in children with osteosarcoma: implications for dosing. Clin Cancer Res. 2014 May 15;20(10):2783-92. doi: 10.1158/1078-0432.CCR-13-2364. Epub 2014 Mar 17. PMID 24637635
- See also: St. Jude Children's Research Hospital — http://www.stjude.org
- See also: Clinical Trials Open at St. Jude — http://www.stjude.org/protocols

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Forty-three participants were enrolled between June 2008 and May 2012: 34 at St. Jude Children's Research Hospital, 6 at Rady Children's Hospital San Diego, 2 at Johns Hopkins University Hospital, and 1 at M.D. Anderson in Houston
Pre-assignment Details: All participants had newly diagnosed high-grade, biopsy-proven osteosarcoma, or malignant fibrous histiocytoma (MFH) of bone
Groups:
- A: Localized Resectable Disease: Stratum A participants had primary tumors potentially resectable by aggressive surgery, such as limb-salvage surgery or amputation, and no evidence of metastasis.
- B: Localized Unresectable Disease: Participants with localized unresectable primary tumors were to participate in Stratum B. No participants were enrolled to this stratum.
- C: Metastatic Tumors: Stratum C participants had metastatic tumors.
Period: Overall Study
Arm/Group | A: Localized Resectable Disease | B: Localized Unresectable Disease | C: Metastatic Tumors
Started | 31 | 0 | 12
Completed | 17 | 0 | 3
Not Completed | 14 | 0 | 9
Not completed — Protocol Violation | 1 | 0 | 0
Not completed — Withdrawal by Subject | 1 | 0 | 0
Not completed — Physician Decision | 3 | 0 | 0
Not completed — Relapse or tumor progression | 9 | 0 | 7
Not completed — Adverse Event | 0 | 0 | 1
Not completed — Ineligible | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Population: Participants were eligible if they were ≤30 years of age on date of diagnostic biopsy confirmation of high-grade osteosarcoma or malignant fibrous histiocytoma (MFH) of bone. Participants had no previous chemotherapy or radiation therapy.
Groups:
- Total: Total of all reporting groups
Arm/Group | A: Localized Resectable Disease | B: Localized Unresectable Disease | C: Metastatic Tumors | Total
Number analyzed (Participants) | 31 | 0 | 12 | 43
Age, Continuous [Mean (Standard Deviation); unit: years] | 12.7 (3.5) |  | 13.3 (4.2) | 12.9 (3.6)
Age, Continuous [Median (Full Range); unit: years] | 12 [6 to 20] |  | 12 [8 to 20] | 12 [6 to 20]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 15 |  | 5 | 20
  Male | 16 |  | 7 | 23

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Unacceptable Toxicity
Description: Objective: To study the feasibility of combining: 1) bevacizumab with cisplatin, doxorubicin, and high-dose methotrexate (MAP) in patients with localized resectable osteosarcoma; and 2) bevacizumab with MAP and ifosfamide, and etoposide in patients with unresectable or metastatic osteosarcoma.
  The target unacceptable toxicity is defined as grade 4 hypertension, proteinuria, or bleeding excluding petechiae/purpura, grade 3/4 thrombosis/embolism excluding catheter-related thrombosis. The unacceptable toxicity for major wound complication is defined as grade 2, 3, or 4 major wound complications.
  A six-stage group sequential stopping rule was developed for monitoring unacceptable toxicity.
Time Frame: After all patients have completed therapy, up to 1 year after last patient is enrolled
Population: Due to slow accrual, the trial was closed to accrual early. Thus, only 31 stratum A patients and 12 stratum B or C patients were enrolled on the study. Therefore, based on the number of patients enrolled and the designed power for the study, we do not have confidence in making a conclusion regarding this feasibility objective.
Measure: Number; unit: participants
Arm/Group | A: Localized Resectable Disease | C: Metastatic Tumors
Number analyzed (Participants) | 31 | 11
participants
  Grade 4 Hypertension | 0 | 0
  Grade 4 Proteinuria | 0 | 0
  Grade 4 Bleeding | 0 | 0
  Grade 3/4 Thrombosis/Embolism | 1 | 0
  Grade 2, 3 or 4 Major Wound Complication | 7 | 2

2. Primary Outcome: 3-Year Event Free Survival
Description: To study the effect of adding bevacizumab to chemotherapy comprised of cisplatin, doxorubicin, and high-dose methotrexate (HDMTX) on the event-free survival (EFS) in patients with localized resectable osteosarcoma. The Kaplan-Meier (K-M) method was used to estimate survival rate.
Time Frame: After all patients have completed therapy, up to 4 years after last patient is enrolled
Measure: Number (95% Confidence Interval); unit: Probability
Groups:
- A: Localized Resectable Disease: OS2008 Stratum A participants had primary tumors potentially resectable by aggressive surgery, such as limb-salvage surgery or amputation, and no evidence of metastasis.
Arm/Group | A: Localized Resectable Disease
Number analyzed (Participants) | 31
Probability | 0.575 [0.402 to 0.747]

3. Secondary Outcome: Histologic Response by Stratum
Description: The effect of adding bevacizumab to preoperative chemotherapy comprised of cisplatin, doxorubicin, and HDMTX on the histologic response in patients with localized resectable osteosarcoma compared to historical controls treated with preoperative cisplatin, doxorubicin, and HDMTX without bevacizumab on the Intergroup Study 0133.
  Histologic response at week 10 of therapy was evaluated by Huvos grading systems as grade I: tumor not responding to therapy, no effect identified; grade IIA: more than 50% viable tumor left; grade IIB: 5-50% viable tumor remaining; grade III: only scattered foci of viable tumor seen (less than 5% of tumor); grade IV: no viable tumor seen in extensive sampling (at least a full cross-section of the tumor).
  The study did not enroll an adequate number of participants, therefore, the comparison to Intergroup Study 0133 participants was not done.
Time Frame: After 6 cycles of chemotherapy, up to 1 year after the start of therapy
Population: All Stratum A participants were evaluated. The tumor sample for analysis was not obtained for one of the 12 Stratum C participants.
Measure: Number; unit: participants
Arm/Group | A: Localized Resectable Disease | C: Metastatic Tumors
Number analyzed (Participants) | 31 | 11
participants
  Grade I | 1 | 0
  Grade IIA | 5 | 1
  Grade IIB | 17 | 7
  Grade III | 8 | 3

4. Secondary Outcome: 2-Year Event Free Survival (EFS) of Patients With Osteosarcoma
Description: Kaplan-Meier method was used to estimate the EFS of patients with osteosarcoma treated with chemotherapy and Bevacizumab.
Time Frame: After all patients have completed therapy, up to 2 years after last patient is enrolled
Population: All the 42 evaluable participants were included in this analysis.
Measure: Number (95% Confidence Interval); unit: probability
Groups:
- All Participants: All the 42 evaluable participants in this study had osteosarcoma, of which 22 had events and 20 had no event.
Arm/Group | All Participants
Number analyzed (Participants) | 42
probability | 0.617 [0.470 to 0.764]

5. Secondary Outcome: 2-Year Overall Survival (OS) of Patients With Osteosarcoma
Description: Kaplan-Meier method was used to estimate the OS of patients with osteosarcoma treated with chemotherapy and Bevacizumab.
Time Frame: After all patients have completed therapy, up to 2 years after last patient is enrolled
Population: All the 42 evaluable participants in this study had osteosarcoma, of which 12 died and 20 were still alive as of 05/04/2015.
Measure: Number (95% Confidence Interval); unit: probability
Groups:
- All Participants: All 42 evaluable participants were included in this analysis
Arm/Group | All Participants
Number analyzed (Participants) | 42
probability | 0.880 [0.782 to 0.978]

6. Secondary Outcome: 2-Year Event Free Survival (EFS) in Patients With Localized Resectable Disease Compared to St. Jude OS99 Protocol.
Description: The current protocol OS2008 (NCT00667342) was closed early due to slow accrual. Thus, with the limited number of patients, the comparison of EFS of OS20008 to that of OS99 (NCT00145639) participants was not done. The 2-year EFS of OS2008 participants is reported here.
Time Frame: After all patients have completed therapy, up to 2 years after last patient is enrolled
Population: OS2008 Localized Resectable Disease group had 31 participants: 14 had events, 17 had no events.
Measure: Number (95% Confidence Interval); unit: probability
Arm/Group | A: Localized Resectable Disease
Number analyzed (Participants) | 31
probability | 0.642 [0.473 to 0.810]

7. Secondary Outcome: 2-Year Overall Survival (OS) in Patients With Localized Resectable Disease Compared to OS99 Protocol.
Description: The current protocol OS2008 (NCT00667342) was closed early due to slow accrual. Thus, with the limited number of patients, the comparison of EFS of OS2008 to that of OS99 (NCT00145639) participants was not done. The 2-year OS of OS2008 participants is reported here.
Time Frame: After all patients have completed therapy, up to 2 years after last patient is enrolled
Population: OS2008 Localized Resectable Disease group had 31 participants: 7 were expired and 24 still alive
Measure: Number (95% Confidence Interval); unit: probability
Arm/Group | A: Localized Resectable Disease
Number analyzed (Participants) | 31
probability | 0.934 [0.847 to 1.0]

8. Secondary Outcome: Mean Ktrans
Description: The volume transfer constant (Ktrans) was used to evaluate clinical outcomes. The average for the distribution across the whole region of interest (ROI) was calculated as a summary measure for each data set.
Time Frame: Baseline through Week 10
Population: The number analyzed at each time point differed due to missing observations at some of the time points
Measure: Mean (Standard Deviation); unit: min(-1)
Arm/Group | A: Localized Resectable Disease | C: Metastatic Tumors
Number analyzed (Participants) | 31 | 11
min(-1)
  Baseline: number analyzed (Participants) | 26 | 9
  Baseline | 0.13 (0.04) | 0.15 (0.07)
  Day -2: number analyzed (Participants) | 21 | 6
  Day -2 | 0.11 (0.05) | 0.14 (0.03)
  Day 1: number analyzed (Participants) | 21 | 6
  Day 1 | 0.12 (0.06) | 0.16 (0.04)
  Day 5: number analyzed (Participants) | 24 | 8
  Day 5 | 0.14 (0.06) | 0.16 (0.04)
  Week 5: number analyzed (Participants) | 28 | 11
  Week 5 | 0.08 (0.04) | 0.10 (0.05)
  Week 10: number analyzed (Participants) | 27 | 11
  Week 10 | 0.07 (0.05) | 0.07 (0.03)
Statistical Analysis 1: Comparison: A: Localized Resectable Disease; Test type: Other — The association between response and Ktrans at Week 10 was evaluated; p = 0.0863, Logistic Regression

9. Secondary Outcome: Mean Vp
Description: The fractional blood plasma volume (Vp) was used to evaluate clinical outcomes. The average for the distribution across the whole region of interest (ROI) was calculated as a summary measure for each data set.
Time Frame: Baseline through Week 10
Population: The number analyzed at each time point differed due to missing observations at some of the time points
Measure: Mean (Standard Deviation); unit: (unitless)
Arm/Group | A: Localized Resectable Disease | C: Metastatic Tumors
Number analyzed (Participants) | 31 | 11
(unitless)
  Baseline: number analyzed (Participants) | 26 | 9
  Baseline | 0.0081 (0.0024) | 0.0094 (0.0016)
  Day -2: number analyzed (Participants) | 21 | 6
  Day -2 | 0.0067 (0.0020) | 0.0077 (0.0022)
  Day 1: number analyzed (Participants) | 21 | 6
  Day 1 | 0.0070 (0.0027) | 0.0095 (0.0027)
  Day 5: number analyzed (Participants) | 24 | 8
  Day 5 | 0.0066 (0.0033) | 0.0089 (0.0029)
  Week 5: number analyzed (Participants) | 28 | 11
  Week 5 | 0.0063 (0.0029) | 0.0069 (0.0032)
  Week 10: number analyzed (Participants) | 27 | 11
  Week 10 | 0.0060 (0.0044) | 0.0055 (0.0026)
Statistical Analysis 1: Comparison: A: Localized Resectable Disease; Test type: Other — The association between response and Vp at Week 10 was evaluated; p = 0.0573, Logistic Regression

10. Secondary Outcome: Mean Ve
Description: The fractional volume of extravascular extracellular space (Ve) was used to evaluate clinical outcomes. The average for the distribution across the whole region of interest (ROI) was calculated as a summary measure for each data set.
Time Frame: Baseline through Week 10
Population: The number analyzed at each time point differed due to missing observations at some of the time points
Measure: Mean (Standard Deviation); unit: (unitless)
Arm/Group | A: Localized Resectable Disease | C: Metastatic Tumors
Number analyzed (Participants) | 31 | 11
(unitless)
  Baseline: number analyzed (Participants) | 26 | 9
  Baseline | 0.2543 (0.0785) | 0.2671 (0.0888)
  Day -2: number analyzed (Participants) | 21 | 6
  Day -2 | 0.2444 (0.0871) | 0.2623 (0.0781)
  Day 1: number analyzed (Participants) | 21 | 6
  Day 1 | 0.2564 (0.1209) | 0.2602 (0.0447)
  Day 5: number analyzed (Participants) | 24 | 8
  Day 5 | 0.2854 (0.1138) | 0.3126 (0.0727)
  Week 5: number analyzed (Participants) | 28 | 11
  Week 5 | 0.3055 (0.1622) | 0.3105 (0.1425)
  Week 10: number analyzed (Participants) | 27 | 11
  Week 10 | 0.2776 (0.1225) | 0.2726 (0.1596)
Statistical Analysis 1: Comparison: A: Localized Resectable Disease; Test type: Other — The association between response and Ve at Week 10 was evaluated; p = 0.0863, Logistic Regression

11. Secondary Outcome: Histologic Response by Number of Participants
Description: The association of interested variables with response was checked with the Wilcoxon rank-sum test. The response is based on the Huvos grade of histologic response for DCE-MRI comparisons and is defined as good for ≥90% necrosis and poor for less than 90%.
Time Frame: at week 10 after start of therapy
Population: Two Stratum A participants with no histologic response were excluded.
Measure: Count of Participants; unit: Participants
Groups:
- All Participants: All 42 evaluable participants in this study had osteosarcoma. This analysis includes 29 Stratum A participants who had primary tumors potentially resectable by aggressive surgery, such as limb-salvage surgery or amputation, and no evidence of metastasis, and 11 Stratum C participants who had metastatic tumors.
Arm/Group | All Participants
Number analyzed (Participants) | 40
Participants
  Poor Response | 22
  Good Response | 18

12. Secondary Outcome: Ktrans by Good and Poor Response
Description: The response is based on the Huvos grade of histologic response for DCE-MRI comparisons and is defined as good for ≥90% necrosis and poor for less than 90%.
Time Frame: at week 10 after start of therapy
Population: Two Stratum A participants with no histologic response were excluded.
Measure: Mean (Standard Error); unit: min(-1)
Arm/Group | All Participants
Number analyzed (Participants) | 40
min(-1)
  Poor Response | 0.0775 (0.0089)
  Good Response | 0.0491 (0.0053)

13. Secondary Outcome: P95 of Ktrans by Good and Poor Response
Description: The response is based on the Huvos grade of histologic response for DCE-MRI comparisons and is defined as good for ≥90% necrosis and poor for less than 90%. P95 denotes the level of each kinetic parameter exceeding 95% of its values in each tumor.
Time Frame: at week 10 after start of therapy
Population: Two Stratum A participants with no histologic response were excluded.
Measure: Mean (Standard Error); unit: min(-1)
Arm/Group | All Participants
Number analyzed (Participants) | 40
min(-1)
  Poor Response | 0.2047 (0.0224)
  Good Response | 0.1228 (0.0136)

14. Secondary Outcome: Difference Between Good and Poor Response by SUVmax
Description: as for outcome 12
Time Frame: at week 10 after start of therapy
Population: One participant with no histologic response but with evaluable imaging was excluded.
Measure: Mean (Standard Error); unit: (unitless)
Groups:
- All Participants: Thirty-two participants with osteosarcoma were evaluated in this study. The analysis for this outcome measure included 23 Stratum A participants who had primary tumors potentially resectable by aggressive surgery, such as limb-salvage surgery or amputation, and no evidence of metastasis, and 8 Stratum C participants who had metastatic tumors.
Arm/Group | All Participants
Number analyzed (Participants) | 31
(unitless)
  Poor Response | 6.2894 (0.9303)
  Good Response | 3.2720 (0.3814)

15. Other Pre Specified Outcome: Number of Participants With Neuropathic Pain (NP) Following Surgery
Description: Of the 43 participants enrolled on this trial, 37 met criteria for evaluation of neuropathic pain (NP) following definitive surgery. The 37 participants underwent 38 surgeries: one participant had a limb-sparing surgery followed by an amputation surgery. Six of 43 participants were excluded from evaluation for NP: 1 due to deep vein thrombosis, 2 removed from study prior to surgery, 1 removed immediately after surgery to receive radiation therapy, 1 had non-extremity osteosarcoma, and 1 patient had a fibula resection. Patients were followed for neuropathic pain daily for the first week postoperatively and weekly for up to 6 months postoperatively.
Time Frame: Up to 6 months postoperatively
Measure: Number; unit: participants
Units Other Than Participants: Number of Surgeries
Groups:
- Amputation Group: Participants had metastatic disease at diagnosis.
- Limb Sparing Group: Participants had localized disease at diagnosis. One participant had 2 surgeries.
- Entire Study Group: Participants enrolled on the study who met the criteria for evaluation of neuropathic pain.
Arm/Group | Amputation Group | Limb Sparing Group | Entire Study Group
Number analyzed (Participants) | 11 | 26 | 37
Number analyzed (Number of Surgeries) | 11 | 27 | 38
participants | 10 | 20 | 30

16. Other Pre Specified Outcome: Median Duration of Neuropathic Pain
Description: Thirty participants who underwent surgery (31 surgeries) were determined to have neuropathic pain. Four participants received only opioids for NP and 26 participants (for 27 surgeries) were treated with NP specific medications including gabapentin, tricyclic antidepressant, methadone. One participant had 2 different surgical procedures and was analyzed both in the limb sparing group and in the amputation group.
Time Frame: From surgery until resolution of NP symptoms, up to 6 months
Population: All participants who met the criteria, had definitive surgery (either limb sparing or/and amputation), experienced neuropathic pain (NP) and were treated for NP until resolution of NP symptoms and off NP medications.
Measure: Median (Full Range); unit: Weeks
Units Other Than Participants: Number of Surgeries
Arm/Group | Amputation Group | Limb Sparing Group | Entire Study Group
Number analyzed (Participants) | 10 | 20 | 30
Number analyzed (Number of Surgeries) | 10 | 21 | 31
Weeks | 3.5 [0.9 to 12.9] | 4.9 [0.3 to 29.9] | 4.4 [0.3 to 29.9]

17. Other Pre Specified Outcome: Mean Duration of Neuropathic Pain
Description: Thirty participants who underwent surgery (31 surgeries) were determined to have neuropathic pain (NP). Four participants received only opioids for NP and 26 participants (for 27 surgeries) were treated with NP specific medications including gabapentin, tricyclic antidepressant, methadone. One participant had 2 different surgical procedures and was analyzed both in the limb sparing group and in the amputation group.
Time Frame: From surgery until resolution of NP symptoms, up to 6 months
Population: All participants who met the criteria, had surgery, experienced neuropathic pain and were treated with NP medication.
Measure: Mean (Standard Deviation); unit: Weeks
Units Other Than Participants: Number of Surgeries
Arm/Group | Amputation Group | Limb Sparing Group | Entire Study Group
Number analyzed (Participants) | 10 | 20 | 30
Number analyzed (Number of Surgeries) | 10 | 21 | 31
Weeks | 4.9 (4.0) | 7.2 (8.4) | 6.5 (7.2)

18. Other Pre Specified Outcome: Median Duration of Neuropathic Pain Medication
Description: as for outcome 17
Time Frame: From surgery until resolution of NP symptoms, up to 6 months
Population: All participants who met the criteria, had surgery, experienced neuropathic pain and were treated with NP medication.
Measure: Median (Full Range); unit: Weeks
Units Other Than Participants: Number of Surgeries
Arm/Group | Amputation Group | Limb Sparing Group | Entire Study Group
Number analyzed (Participants) | 10 | 16 | 26
Number analyzed (Number of Surgeries) | 10 | 17 | 27
Weeks | 6.5 [3.0 to 30.0] | 7.0 [1.7 to 29.9] | 7.0 [1.7 to 30.0]

19. Other Pre Specified Outcome: Mean Duration of Neuropathic Pain Medication
Description: as for outcome 16
Time Frame: From surgery until resolution of NP symptoms, up to 6 months
Measure: Mean (Standard Deviation); unit: Weeks
Units Other Than Participants: Number of Surgeries
Arm/Group | Amputation Group | Limb Sparing Group | Entire Study Group
Number analyzed (Participants) | 10 | 16 | 26
Number analyzed (Number of Surgeries) | 10 | 17 | 27
Weeks | 9.0 (8.0) | 9.8 (8.4) | 9.5 (8.1)

ADVERSE EVENTS:
Time Frame: Adverse events were recorded from on-study date through April 2015.
Arm/Group | A: Localized Resectable Disease | C: Metastatic Tumors
Serious Adverse Events (participants affected / at risk) | 3/31 | 0/11
Other Adverse Events (participants affected / at risk) | 31/31 | 11/11
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | A: Localized Resectable Disease (N=31) | C: Metastatic Tumors (N=11)
Hypotension (Cardiac disorders) | 1 (1) | 0 (0)
Fever (in the absence of neutropenia, where neutropenia is defined as ANC <1.0 x 10e9/L) (General disorders) | 1 (1) | 0 (0)
Infection with normal ANC or Grade 1 or 2 neutrophils, Lung (pneumonia) (Infections and infestations) | 1 (1) | 0 (0)
Cognitive disturbance (Nervous system disorders) | 1 (1) | 0 (0)
Encephalopathy (Nervous system disorders) | 1 (1) | 0 (0)
Neuropathy: motor (Nervous system disorders) | 1 (1) | 0
Neuropathy: sensory (Nervous system disorders) | 1 (1) | 0 (0)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | A: Localized Resectable Disease (N=31) | C: Metastatic Tumors (N=11)
ALT, SGPT (serum glutamic pyruvic transaminase) (Metabolism and nutrition disorders) | 29 (291) | 10 (90)
Albumin, serum-low (hypoalbuminemia) (Metabolism and nutrition disorders) | 29 (258) | 10 (90)
Hemoglobin (Blood and lymphatic system disorders) | 30 (255) | 11 (135)
Leukocytes (total WBC) (Blood and lymphatic system disorders) | 30 (230) | 11 (123)
Platelets (Blood and lymphatic system disorders) | 30 (212) | 11 (137)
AST, SGOT (serum glutamic oxaloacetic transaminase) (Metabolism and nutrition disorders) | 29 (296) | 10 (91)
Glucose, serum-high (hyperglycemia) (Metabolism and nutrition disorders) | 13 (75) | 5 (21)
Phosphate, serum-low (hypophosphatemia) (Metabolism and nutrition disorders) | 26 (144) | 9 (71)
Mucositis/stomatitis (clinical exam), oral cavity (Gastrointestinal disorders) | 25 (101) | 7 (39)
Nausea (Gastrointestinal disorders) | 24 (173) | 7 (65)
Vomiting (Gastrointestinal disorders) | 25 (148) | 8 (47)
Hemorrhage, pulmonary/upper respiratory, Nose (Respiratory, thoracic and mediastinal disorders) | 23 (106) | 9 (38)
Sodium, serum-low (hyponatremia) (Metabolism and nutrition disorders) | 23 (128) | 6 (43)
Proteinuria (Metabolism and nutrition disorders) | 20 (69) | 11 (42)
Anorexia (Gastrointestinal disorders) | 22 (84) | 8 (30)
Potassium, serum-low (hypokalemia) (Metabolism and nutrition disorders) | 21 (146) | 10 (73)
Calcium, serum-low (hypocalcemia) (Metabolism and nutrition disorders) | 20 (80) | 7 (20)
Febrile neutropenia (Infections and infestations) | 20 (34) | 8 (18) — Fever of unknown origin without clinically or microbiologically documented infection) (ANC <1.0 x 10e9/L)
Pain, Abdomen NOS (General disorders) | 15 (43) | 4 (9)
Weight loss (General disorders) | 19 (112) | 7 (36)
Bilirubin (hyperbilirubinemia) (Metabolism and nutrition disorders) | 18 (98) | 6 (17)
Pain, Head/headache (General disorders) | 16 (45) | 6 (9)
Constipation (Gastrointestinal disorders) | 12 (30) | 4 (10)
Magnesium, serum-low (hypomagnesemia) (Metabolism and nutrition disorders) | 16 (105) | 6 (34)
Fever (in the absence of neutropenia, where neutropenia is defined as ANC <1.0 x 10e9/L) (General disorders) | 14 (43) | 2 (3)
Allergic rhinitis (including sneezing, nasal stuffiness, postnasal drip) (Immune system disorders) | 6 (8) | 2 (2)
Pain, extremity-limb (General disorders) | 4 (6) | 0 (0)
Hypertension (Cardiac disorders) | 12 (29) | 1 (1)
Rash/desquamation (Skin and subcutaneous tissue disorders) | 12 (23) | 2 (2)
Allergic reaction/hypersensitivity (including drug fever) (Immune system disorders) | 5 (6) | 1 (1)
Fatigue (asthenia, lethargy, malaise) (General disorders) | 13 (40) | 4 (17)
Diarrhea (Gastrointestinal disorders) | 13 (31) | 3 (7)
Hearing: patients with/without baseline audiogram and enrolled in a monitoring program (Ear and labyrinth disorders) | 14 (19) | 6 (11)
Pain, oral cavity (General disorders) | 14 (28) | 6 (13)
Pain, throat/pharynx/larynx (General disorders) | 12 (28) | 5 (11)
Supraventricular and nodal arrhythmia, sinus tachycardia (Cardiac disorders) | 9 (14) | 2 (3)
Cough (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 0 (0)
Uric acid, serum-high (hyperuricemia) (Metabolism and nutrition disorders) | 8 (19) | 1 (1)
Pruritus/itching (Skin and subcutaneous tissue disorders) | 5 (5) | 2 (3)
Pain, Back (General disorders) | 3 (3) | 0 (0)
Dizziness (Nervous system disorders) | 5 (5) | 3 (4)
Glucose, serum-low (hypoglycemia) (Metabolism and nutrition disorders) | 2 (2) | 1 (2)
Hair loss/alopecia (scalp or body) (Skin and subcutaneous tissue disorders) | 9 (11) | 3 (3)
Dehydration (Gastrointestinal disorders) | 8 (9) | 3 (4)
Pain, chest/thorax NOS (General disorders) | 4 (7) | 0 (0)
Hemoglobinuria (Metabolism and nutrition disorders) | 7 (8) | 0 (0)
Potassium, serum-high (hyperkalemia) (Metabolism and nutrition disorders) | 3 (4) | 1 (1)
Bicarbonate, serum-low (Metabolism and nutrition disorders) | 8 (24) | 4 (8)
Magnesium, serum-high (hypermagnesemia) (Metabolism and nutrition disorders) | 7 (13) | 2 (3)
Hemorrhage, GI, rectum (Gastrointestinal disorders) | 4 (4) | 3 (5)
GGT (gamma-glutamyl transpeptidase) (Metabolism and nutrition disorders) | 5 (24) | 4 (14)
Mucositis/stomatitis (functional/symptomatic), oral cavity (Gastrointestinal disorders) | 7 (11) | 6 (9)
Urinary retention (including neurogenic bladder) (Renal and urinary disorders) | 2 (2) | 0 (0)
Lymphopenia (Blood and lymphatic system disorders) | 6 (31) | 1 (5)
Heartburn/dyspepsia (Gastrointestinal disorders) | 4 (6) | 0 (0)
Sodium, serum-high (hypernatremia) (Metabolism and nutrition disorders) | 4 (4) | 1 (1)
Tinnitus (Ear and labyrinth disorders) | 6 (8) | 1 (2)
Neuropathy: sensory (Nervous system disorders) | 3 (4) | 0 (0)
Creatinine (Metabolism and nutrition disorders) | 6 (11) | 4 (6)
Skin breakdown/decubitus ulcer (Skin and subcutaneous tissue disorders) | 2 (3) | 0 (0)
Calcium, serum-high (hypercalcemia) (Metabolism and nutrition disorders) | 3 (3) | 0 (0)
Prolonged QTc interval (Cardiac disorders) | 5 (7) | 1 (1)
Infection with normal ANC or Grade 1 or 2 neutrophils, skin (cellulitis) (Infections and infestations) | 3 (3) | 0 (0)
Hypotension (Cardiac disorders) | 3 (4) | 1 (1)
Pain, esophagus (General disorders) | 5 (14) | 2 (2)
Hemorrhage, GU, bladder (Renal and urinary disorders) | 3 (5) | 2 (2)
Alkaline phosphatase (Metabolism and nutrition disorders) | 5 (14) | 3 (4)
Left ventricular systolic dysfunction (Cardiac disorders) | 8 (12) | 5 (7)
Hemorrhage, GI, lower GI NOS (Gastrointestinal disorders) | 4 (6) | 0 (0)
Pain, urethra (General disorders) | 2 (2) | 0 (0)
Esophagitis (Gastrointestinal disorders) | 4 (6) | 1 (1)
Hemorrhage, GI, upper GI NOS (Gastrointestinal disorders) | 4 (4) | 1 (1)
Hemorrhage, GU, urinary NOS (Renal and urinary disorders) | 3 (3) | 1 (1)
Pain, joint (General disorders) | 2 (4) | 0 (0)
Pain, phantom (pain associated with missing limb) (General disorders) | 2 (2) | 1 (1)
Mucositis/stomatitis (functional/symptomatic), esophagus (Gastrointestinal disorders) | 4 (4) | 2 (2)
Infection with normal ANC or Grade 1 or 2 neutrophils, catheter-related (Infections and infestations) | 3 (4) | 1 (2)
Glomerular filtration rate (Metabolism and nutrition disorders) | 4 (4) | 2 (2)
Vision-blurred vision (Eye disorders) | 2 (2) | 0 (0)
Pain, rectum (General disorders) | 3 (6) | 2 (3)
Chelitis (Skin and subcutaneous tissue disorders) | 4 (5) | 1 (1)
Fracture (Musculoskeletal and connective tissue disorders) | 2 (3) | 1 (1)
Urinary electrolyte wasting (e.g., Fanconi's syndrome, renal tubular acidosis) (Renal and urinary disorders) | 3 (3) | 5 (7)
Neutrophils/granulocytes (ANC/AGC) (Blood and lymphatic system disorders) | 31 (241) | 11 (130)
Conduction abnormality/atrioventricular heart block, conduction abnormality, NOS (Cardiac disorders) | 2 (2) | 0 (0)
Mucositis/stomatitis (clinical exam), anus (Gastrointestinal disorders) | 3 (5) | 0 (0)
Hemorrhage, GI, anus (Gastrointestinal disorders) | 2 (2) | 0 (0)
Infection with normal ANC or Grade 1 or 2 neutrophils, blood (Infections and infestations) | 2 (2) | 0 (0)
Pain, stomach (General disorders) | 2 (2) | 0 (0)
Infection with Grade 3 or 4 neutrophils (ANC <1.0 x 10e9/L), skin (cellulitis) (Infections and infestations) | 2 (2) | 1 (1) — Documented clinically or microbiologically
Confusion (Psychiatric disorders) | 2 (2) | 0 (0)
Irregular menses (change from baseline) (Reproductive system and breast disorders) | 3 (4) | 1 (2)
Pain, pain NOS (General disorders) | 3 (6) | 1 (1)
Hemorrhage, GI, oral cavity (Gastrointestinal disorders) | 2 (4) | 2 (2)
Infection with normal ANC or Grade 1 or 2 neutrophils, oral cavity-gums (gingivitis) (Infections and infestations) | 3 (6) | 2 (4)
Rigors/chills (General disorders) | 2 (2) | 0 (0)
Colitis, infectious (e.g., Clostridium difficile) (Infections and infestations) | 2 (3) | 0 (0)
Infection with normal ANC or Grade 1 or 2 neutrophils, wound (Infections and infestations) | 2 (2) | 0 (0)
Encephalopathy (Nervous system disorders) | 2 (2) | 0 (0)
Pulmonary/upper respiratory - other (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0)
Pain, pleura (General disorders) | 2 (5) | 0 (0)
Mucositis/stomatitis (clinical exam), esophagus (Gastrointestinal disorders) | 2 (2) | 1 (1)
Mucositis/stomatitis (clinical exam), rectum (Gastrointestinal disorders) | 2 (2) | 1 (1)
Taste alteration (dysgeusia) (Gastrointestinal disorders) | 2 (2) | 0 (0)
Hemorrhage, pulmonary/upper respiratory, bronchopulmonary NOS (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Infection with Grade 3 or 4 neutrophils (ANC <1.0 x 10e9/L), blood (Infections and infestations) | 2 (2) | 1 (1) — Documented clinically or microbiologically.
Joint-effusion (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Infection with Grade 3 or 4 neutrophils (ANC <1.0 x 10e9/L), oral cavity-gums (Infections and infestations) | 2 (3) | 2 (2) — Documented clinically or microbiologically.
Somnolence/depressed level of consciousness (Nervous system disorders) | 0 (0) | 1 (1)
Infection with normal ANC or Grade 1 or 2 neutrophils, mucosa (Infections and infestations) | 2 (2) | 3 (3)
Neuropathy: motor (Nervous system disorders) | 1 (1) | 2 (2)
Infection with Grade 3 or 4 neutrophils (ANC <1.0 x 10e9/L), catheter-related (Infections and infestations) | 2 (2) | 5 (7) — Documented clinically or microbiologically.
Rash: hand-foot skin reaction (Skin and subcutaneous tissue disorders) | 1 (2) | 1 (1)
Mucositis/stomatitis (functional/symptomatic), pharynx (Gastrointestinal disorders) | 1 (1) | 1 (1)
Proctitis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Bone age (alteration in bone age) (General disorders) | 1 (1) | 1 (1)
Infection with Grade 3 or 4 neutrophils (ANC <1.0 x 10e9/L), lung (pneumonia) (Infections and infestations) | 1 (1) | 1 (1) — Documented clinically or microbiologically.
Infection with normal ANC or Grade 1 or 2 neutrophils, bladder (urinary) (Infections and infestations) | 0 (0) | 1 (1)
Infection with normal ANC or Grade 1 or 2 neutrophils, urinary tract NOS (Infections and infestations) | 0 (0) | 1 (1)
Pain, anus (General disorders) | 1 (1) | 1 (1)
Hemorrhage/bleeding - other (General disorders) | 1 (1) | 2 (2)
Supraventricular and nodal arrhythmia, sinus arrhythmia (Cardiac disorders) | 0 (0) | 1 (1)
Injection site reaction/extravasation changes (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Infection with Grade 3 or 4 neutrophils (ANC <1.0 x 10e9/L), conjunctiva (Infections and infestations) | 0 (0) | 1 (1) — Documented clinically or microbiologically)
Infection with Grade 3 or 4 neutrophils (ANC <1.0 x 10e9/L), eye NOS (Infections and infestations) | 0 (0) | 1 (1)
Infection with Grade 3 or 4 neutrophils (ANC <1.0 x 10e9/L), mucosa (Infections and infestations) | 0 (0) | 1 (1) — Documented clinically or microbiologically.
Infection with Grade 3 or 4 neutrophils (ANC <1.0 x 10e9/L), urinary tract NOS (Infections and infestations) | 0 (0) | 1 (1) — Documented clinically or microbiologically.
Infection with normal ANC or Grade 1 or 2 neutrophils, lung (pneumonia) (Infections and infestations) | 0 (0) | 1 (1)
Pain, lip (General disorders) | 0 (0) | 1 (1)
Infection (ANC <1.0 x 10e9/L, fever >38.5 degrees C.), blood (Infections and infestations) | 0 (0) | 2 (2) — Documented clinically or microbiologically.
Infection with normal ANC or Grade 1 or 2 neutrophils, colon (Infections and infestations) | 0 (0) | 2 (3)

LIMITATIONS AND CAVEATS:
Accrual to this study was stopped early after 4.5 years due to slow accrual of participants. No eligible participants were enrolled on Stratum B. All enrolled participants continue on study and results will be reported when available.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes